CLINICAL TRIAL: NCT05203289
Title: Relative Bioavailability of 40 mg/0.4 mL of BI 695501 Compared to 40 mg/0.8 mL of BI 695501 Formulation Following Single Subcutaneous Administration in Healthy Male and Female Subjects (a Double Blind, Randomised, Single-dose, Parallel-arm Study)
Brief Title: A Study in Healthy People to Test How 2 Different Formulations of BI 695501 Are Taken up by the Body When Given as an Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1297-0015
Record Dates: First submitted 2022-01-13; First posted 2022-01-24 (Actual); Results first posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2023-08

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BI 695501 40 mg/0.4 mL (T) (Experimental): Participants were subcutaneously injected 40 milligram (mg)/0.4 milliliter (mL) of BI 695501 solution for injection in prefilled syringe (PFS) (Test Treatment (T)).
  Interventions: Drug: BI 695501 - higher concentration
- BI 695501 40 mg/0.8 mL (R) (Experimental): Participants were subcutaneously injected 40 milligrams (mg)/0.8 milliliter (mL) of BI 695501 solution for injection in prefilled syringe (PFS) (Reference Treatment (R)).
  Interventions: Drug: BI 695501 - lower concentration

INTERVENTIONS:
Drug: BI 695501 - higher concentration — BI 695501 - higher concentration
  Arms: BI 695501 40 mg/0.4 mL (T)
Drug: BI 695501 - lower concentration — BI 695501 - lower concentration
  Arms: BI 695501 40 mg/0.8 mL (R)

SUMMARY:
The main objective of this trial is to compare the pharmacokinetics (PK) of 40 mg BI 695501 100 mg/mL with 40 mg BI 695501 50 mg/mL following single subcutaneous administration.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects according to the assessment of the investigator, as based on a complete medical history including a physical examination, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests.
* Age of 18 to 55 years (inclusive).
* Body mass index (BMI) of 18.5 to 29.9 kg/m2 (inclusive).
* Signed and dated written informed consent in accordance with International Council for Harmonisation-Good Clinical Practice (ICH-GCP) and local legislation prior to admission to the trial.
* Participants of reproductive potential (childbearing potential1) must be willing and able to use highly effective methods of birth control per International Council for Harmonisation (ICH) M3 (R2) that result in a low failure rate of less than 1% per year from at least 30 days before administration of the trial medication until 30 days after trial completion.

Exclusion Criteria:

* Previous exposure to adalimumab or proposed adalimumab biosimilar drugs.
* Any finding in the medical examination (including blood pressure (BP), pulse rate (PR) or electrocardiogram (ECG)) that deviates from normal and judged as clinically relevant by the investigator.
* Any evidence of a concomitant disease judged as clinically relevant by the investigator including gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological, hormonal disorders or diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders.
* History of relevant orthostatic hypotension, fainting spells, or blackouts.
* Chronic or relevant acute infections.
* Positive result for human immunodeficiency virus (HIV), hepatitis B virus (HBV), and hepatitis C (Hep C) at screening.
* History of relevant allergy or hypersensitivity including allergy to the trial medication, its excipients or device materials (e.g. natural rubber or latex).
* Within 10 days prior to administration of trial medication, use of drugs that might reasonably influence the results of the trial.

Further exclusion criteria apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2022-02-18 (Actual); Primary Completion 2022-08-29 (Actual); Study Completion 2022-08-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Miami Research Associates, Inc, Miami, Florida
  - QPS MO, Springfield, Missouri

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Moschetti V, Buschke S, Bertulis J, Hohl K, McCabe D. Relative bioavailability, immunogenicity, and safety of two adalimumab-adbm formulations in healthy volunteers: a double-blind, randomized, single-dose, parallel-arm Phase I trial (VOLTAIRE-HCLF). Expert Opin Biol Ther. 2024 Jul;24(7):673-679. doi: 10.1080/14712598.2024.2354902. Epub 2024 May 19. PMID 38739422
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 14-week, randomized, single dose, parallel arm, double blind, Phase I trial in healthy male and female subjects aged ≥18 to ≤55 years. The aim of this trial was to evaluate and compare the pharmacokinetics (PK), safety, tolerability, and immunogenicity of the test treatment to the reference treatment administered subcutaneously via prefilled syringe (PFS).
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trials. There was no run-in period and subjects did not have to attend a specialist site. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Period: Overall Study
Arm/Group | BI 695501 40 mg/0.4 mL (T) | BI 695501 40 mg/0.8 mL (R)
Started | 99 | 101
Completed (Completed Treatment) | 99 | 101
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects randomized set (RND): All subjects randomized set contained all subjects who provided informed consent for this study (all subjects enrolled set (ENR)) and were randomized to trial medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | BI 695501 40 mg/0.4 mL (T) | BI 695501 40 mg/0.8 mL (R) | Total
Number analyzed (Participants) | 99 | 101 | 200
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.4 (9.82) | 37.5 (8.41) | 37.0 (9.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 47 | 104
  Male | 42 | 54 | 96
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 51 | 55 | 106
  Not Hispanic or Latino | 48 | 46 | 94
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 90 | 93 | 183
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve of BI 695501 in Plasma Over the Time Interval From 0 to 1344 Hours After Dose Administration (AUC0-1344)
Description: Area under the concentration-time curve of BI 695501 in plasma over the time interval from 0 to 1344 hours after dose administration (AUC0-1344).
  The presented means are adjusted based on analysis of covariance (ANCOVA) model on the logarithmic scale with fixed effects for treatment, location of trial medication injection and baseline body weight.
Time Frame: BI 695501 was measured within 1 hour before and 4, 12, 24, 48, 72, 96, 120, 144, 168, 216, 336, 504, 672, 840, 1008 and 1344 hours after drug administration.
Population: Pharmacokinetic analysis set (PKS): The pharmacokinetic set consisted of all randomized subjects who received the single dose of trial medication, and had at least one evaluable primary pharmacokinetics (PK) parameter, and were without important protocol deviations or violations thought to have a relevant impact on the PK of BI 695501.
  Only participants with evaluable results for this PK parameter are reported.
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Microgram * hours / milliliter
Arm/Group | BI 695501 40 mg/0.4 mL (T) | BI 695501 40 mg/0.8 mL (R)
Number analyzed (Participants) | 93 | 99
Microgram * hours / milliliter | 1415.103 (37.600) | 1389.021 (37.600)
Statistical Analysis 1: Comparison: BI 695501 40 mg/0.4 mL (T) vs BI 695501 40 mg/0.8 mL (R); The statistical model used for the analysis of the primary endpoints was an analysis of covariance (ANCOVA) model on the logarithmic scale. The PK endpoints were log-transformed (natural logarithm) prior to fitting the ANCOVA model. This model included effects accounting for the following sources of variation: 'treatment', 'location of trial medication injection' and 'baseline body weight' (continuous); Test type: Other; Ratio of geometric means (%) = 101.88, 90% CI 2-sided [93.31 to 111.23] — The estimated parameter was the adjusted geometric mean ratios (%) of BI 695501: (40 mg/0.4 mL (T))/(40 mg/0.8 mL (R)). Geometric standard error= 105.455

2. Primary Outcome: Area Under the Concentration-time Curve of BI 695501 in Plasma Over the Time Interval From 0 Extrapolated to Infinity (AUC0-∞)
Description: Area under the concentration-time curve of BI 695501 in plasma over the time interval from 0 extrapolated to infinity (AUC0-∞).
  The presented means are adjusted based on analysis of covariance (ANCOVA) model on the logarithmic scale with fixed effects for treatment, location of trial medication injection and baseline body weight.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Microgram * hours / milliliter
Arm/Group | BI 695501 40 mg/0.4 mL (T) | BI 695501 40 mg/0.8 mL (R)
Number analyzed (Participants) | 93 | 99
Microgram * hours / milliliter | 1518.311 (44.690) | 1440.860 (44.690)
Statistical Analysis 1: Comparison: BI 695501 40 mg/0.4 mL (T) vs BI 695501 40 mg/0.8 mL (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of geometric means (%) = 105.38, 90% CI 2-sided [95.06 to 116.81] — The estimated parameter was the adjusted geometric mean ratios (%) of BI 695501: (40 mg/0.4 mL (T))/(40 mg/0.8 mL (R)). Geometric standard error= 106.431

3. Primary Outcome: Maximum Measured Concentration of BI 695501 in Plasma (Cmax)
Description: Maximum measured concentration of BI 695501 in plasma (Cmax). The presented means are adjusted based on analysis of covariance (ANCOVA) model on the logarithmic scale with fixed effects for treatment, location of trial medication injection and baseline body weight.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Least Squares Mean (Geometric Coefficient of Variation); unit: Microgram / milliliter
Arm/Group | BI 695501 40 mg/0.4 mL (T) | BI 695501 40 mg/0.8 mL (R)
Number analyzed (Participants) | 98 | 101
Microgram / milliliter | 2.811 (34.215) | 3.079 (34.215)
Statistical Analysis 1: Comparison: BI 695501 40 mg/0.4 mL (T) vs BI 695501 40 mg/0.8 mL (R); [analysis description as in outcome 1, analysis 1]; Test type: Other; Ratio of geometric means (%) = 91.29, 90% CI 2-sided [84.38 to 98.76] — The estimated parameter was the adjusted geometric mean ratios (%) of BI 695501: (40 mg/0.4 mL (T))/(40 mg/0.8 mL (R)). Geometric standard error= 104.874

ADVERSE EVENTS:
Time Frame: From first drug administration until the end of study (e.o.s.) examination. That means up to 70 days.
Description: Safety analysis set (SAF): The SAF included all subjects who were randomized and treated with study drug and will be analyzed according to treatment received.
Arm/Group | BI 695501 40 mg/0.4 mL (T) | BI 695501 40 mg/0.8 mL (R)
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/101
Serious Adverse Events (participants affected / at risk) | 0/99 | 0/101
Other Adverse Events (participants affected / at risk) | 6/99 | 13/101
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BI 695501 40 mg/0.4 mL (T) (N=99) | BI 695501 40 mg/0.8 mL (R) (N=101)
Injection site erythema (General disorders) | 1 | 8
Headache (Nervous system disorders) | 5 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-11-26): https://cdn.clinicaltrials.gov/large-docs/89/NCT05203289/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-30): https://cdn.clinicaltrials.gov/large-docs/89/NCT05203289/SAP_001.pdf